CLINICAL TRIAL: NCT02850094
Title: The Brigham and Women's Hospital Wellness Project
Brief Title: The BWH Wellness Project
Acronym: B-Well
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elena Losina, Professor of Orthopaedic Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000970
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2016-07

CONDITIONS: Physical Activity
Keywords: Physical activity; Exercise; Financial Incentives
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Financial Bonuses (Experimental): For two weeks following enrollment, subjects are monitored via their FitBit accelerometer to monitor their pre-intervention physical activity levels. For a twenty-four week period following the observational period, participants are eligible for financial bonuses based on their increased activity. Participants enroll as teams and are eligible for additional financial bonuses based on their team's performance.
  Interventions: Behavioral: Financial Bonuses

INTERVENTIONS:
Behavioral: Financial Bonuses — Each participant is eligible to receive $10 per week for increasing their minutes of moderate to vigorous physical activity by 10% from the previous week, or for meeting CDC guidelines of 150 minutes/week. Participants who meet their target minutes of PA every week for one month, three months, or six months receive $15, $25, or $50 bonuses respectively. If all members of a team meet their individual PA goals, each participant's reward is doubled. In total, participants can earn up to $860 if they meet all their goals.

SUMMARY:
The investigators propose a 24 week program to provide proof-of-principle evidence that financial incentives stimulate Brigham and Women's Hospital (BWH) employees to be more physically active.

DETAILED DESCRIPTION:
Participants wear a Fitbit Flex accelerometer for at least six months. During the first two weeks, they are paid simply for wearing the Fitbit. After that, they are regularly paid for either meeting CDC guidelines for moderate physical activity (PA) or increasing their PA by at least 10% from the preceding week. Moderate PA is defined as walking for at least 100 steps per minute for at least 10 minutes at a time. One minute of vigorous PA, over 175 steps/minute, counts as two minutes of moderate PA.

In addition to weekly bonuses, there are also bonuses for achieving all goals in 1 month, 3 month, and 6 month intervals. In cases where all three team members received a bonus, their bonuses are doubled. Individuals also fill out weekly questionnaires about their work attendance, as well as longer questionnaires at baseline, three months, and six months.

ELIGIBILITY:
Inclusion Criteria:

* Brigham and Women's Hospital employee
* Reported less than 30 minutes of exercise per week
* Use a computer daily at work or home
* Willing to wear a pedometer, undergo health screening, and complete occasional questionnaires

Exclusion Criteria:

* Occupation: Physician, nurse or other clinician
* Self-reported pregnancy at baseline

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 6 Months
  Minutes of moderate to vigorous physical activity (greater than 100 steps/minute)

SECONDARY OUTCOMES:
Individuals Meeting CDC Guidelines | 6 Months
  Percentage of cohort that achieved 150 minutes of moderate PA per week
Fitbit Adherence | 6 Months
  Percentage of cohort that wore their Fitbit for four or more days per week for at least 20 out of 24 weeks

REFERENCES:
- [Derived] Meints SM, Yang HY, Collins JE, Katz JN, Losina E. Race Differences in Physical Activity Uptake Within a Workplace Wellness Program: A Comparison of Black and White Employees. Am J Health Promot. 2019 Jul;33(6):886-893. doi: 10.1177/0890117119833341. Epub 2019 Feb 26. PMID 30808208
- [Derived] Losina E, Smith SR, Usiskin IM, Klara KM, Michl GL, Deshpande BR, Yang HY, Smith KC, Collins JE, Katz JN. Implementation of a workplace intervention using financial rewards to promote adherence to physical activity guidelines: a feasibility study. BMC Public Health. 2017 Dec 1;17(1):921. doi: 10.1186/s12889-017-4931-2. PMID 29195494
- [Derived] Smith KC, Michl GL, Katz JN, Losina E. Meteorologic and Geographic Barriers to Physical Activity in a Workplace Wellness Program. J Phys Act Health. 2018 Feb 1;15(2):108-116. doi: 10.1123/jpah.2016-0731. Epub 2017 Nov 25. PMID 28872399